CLINICAL TRIAL: NCT04219722
Title: Treatment of Symptoms Associated With Vulvovaginal Atrophy in Postmenopausal Women by Hyaluronic Acid Injection Into the Vaginal Mucosa
Brief Title: Efficacy and Safety of Hyaluronic Acid Injection on Symptoms of Vulvovaginal Atrophy in Postmenopausal Women
Acronym: SYLIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-A00034-53
Record Dates: First submitted 2019-12-18; First posted 2020-01-07 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Vulvovaginal Atrophy
Keywords: Vaginal dryness; Vulvovaginal symptoms; Hyaluronic acid; Injection; Postmenopause; Prospective; 2-step study; Single-blind; Randomized; Placebo; Open study

STUDY DESIGN:
Intervention Model Description: Study performed in two steps:
  * From 0 to 12 weeks: randomized, single-blind, placebo-controlled study
  * From 12 to 52 weeks: open label, treatment only study
Who Masked: Participant
Masking Description: Subjects will be blinded during the first 12 weeks of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desirial only group (Active Comparator): Administration of DESIRIAL® at Day 0 (Visit 1)
  Interventions: Device: Injection of DESIRIAL®
- Placebo and Desirial group (Placebo Comparator): Administration of placebo at Day 0 (Visit 1). If still eligible 12 weeks (Visit 3) after placebo injection, patient will be treated with DESIRIAL®
  Interventions: Device: Injection of DESIRIAL®; Other: Injection of placebo

INTERVENTIONS:
Device: Injection of DESIRIAL® — DESIRIAL® is a hyaluronic acid injectable gel intended to treat symptoms associated with vulvovaginal atrophy in postmenopausal women by vaginal mucosa rehydration in this study.
  1 mL of DESIRIAL® will be injected in the vestibule and on the posterior and lateral walls of the vagina, 2 to 3 cm after the introitus.
  Other Names: Injection of hyaluronic acid gel
Other: Injection of placebo — Placebo is an isotonic saline solution (0.9% NaCl).
  1 mL of placebo will be injected in the vestibule and on the posterior and lateral walls of the vagina, 2 to 3 cm after the introitus.
  Other Names: Injection of NaCl 0.9%
  Arms: Placebo and Desirial group

SUMMARY:
DESIRIAL® is a CE-marketed hyaluronic acid gel intented to rehydrate vaginal and vestibular mucous membranes by mucosal injections. In this study, 121 postmenopausal women of minimum age 45 with symptoms associated with vulvovaginal atrophy, refusing estrogen therapies for treatment of symptoms or with contraindications for such therapies, with at least one moderate to severe vulvovaginal symptom among dryness sensation, dyspareunia, itching / irritation and pain, who have given her informed consent and met all the eligibility criteria, will be enrolled. Patients will randomly receive 1 injection of DESIRIAL® or placebo (ratio 2:1) in the vaginal mucosa at Day 0. If still eligible 12 weeks after, patients receiving placebo at Day 0 will be treated with DESIRIAL®. Patients will come to a total of 6 to 8 visits depending on the product injected at Day 0 over a period of 11 up to 12 months. Phone interview will be performed between 3 and 5 days after injection. Variation of vulvovaginal symptomatology, sexual function, vaginal pH and safety will be assessed.

DETAILED DESCRIPTION:
This is a prospective, international, multicenter study performed in 2 steps:

* From 0 to 12 weeks: randomized, single-blind, placebo-controlled study;
* From 12 to 52 weeks: open label, treatment only study.

The study will assess the efficacy of DESIRIAL® in reducing the vulvovaginal symptomatology after a single injection. One hundred twenty one postmenopausal women of minimum age 45, with symptoms associated with vulvovaginal atrophy, refusing estrogen therapies for treatment of symptoms or with contraindications for such therapies, with at least one moderate to severe vulvovaginal symptom among dryness sensation, dyspareunia, itching / irritation and pain, who have given her informed consent and met all the eligibility criteria, will be enrolled. Patients will randomly (2:1 ratio) receive a 1mL-injection of DESIRIAL® (Desirial Only group, DO) or placebo (Placebo and Desirial group, PAD) in the vestibular and vaginal mucosa using the multi-puncture and/or retrolinear technique at D0. If still eligible 12 weeks after, patients from PAD group receiving placebo at Day 0 will be treated with DESIRIAL®. Group DO will be followed up at 4, 12, 24, 36 and 52 weeks timepoints.Group PAD will be followed up at 4, 12, 16, 24, 36 and 48 weeks timepoints. Phone interview will be performed between 3 and 5 days after injection to check safety. Variation of vulvovaginal symptomatology, sexual function and vaginal pH will be measured using vulvovaginal symptomatology questionnaire, Female Sexual Function Index (FSFI) and vaginal pH indicator strip respectively. Safety will also be assessed through collection of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 45 years of age at inclusion;
* With postmenopausal status: at least 12 months of spontaneous amenorrhea or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy at the time of inclusion. Hormone-dependent breast cancer survivors previously treated with long-term anti-estrogen treatment tamoxifene, in complete remission of breast cancer, and with a post-menopause diagnosis after tamoxifene discontinuation are eligible;
* Refusing estrogen therapies for treatment of vulvovaginal symptomatology or with contraindications for such therapies;
* With at least one of the following vulvovaginal symptoms, as moderate to severe, self-assessed: Dryness sensation, Dyspareunia, Itching / irritation, Pain. Possible scores are 0 - none, 1 - mild, 2 - moderate, 3 - severe;
* Subject affiliated to a health social security system (if applicable according to national regulation);
* Informed consent signed by the patient for study enrolment.

Exclusion Criteria:

Women with the following conditions:

* General:

  * Pregnancy;
  * Breast feeding;
  * With a known tendency to develop hypertrophic or keloid scars;
  * Participating at the same time in another clinical trial;
  * Deprived of their freedom by administrative or legal decision or under trusteeship/guardianship;
  * With a known and documented hypernatremia;
  * With a known and documented hyperchloremia;
  * With a severe case of hydric inflation and hydro-sodic retention, particularly in case of decompensated heart failure, decompensated liver failure (cirrhosis with oedema and ascites), and pre-eclampsia / eclampsia.
* Linked to genital status: With a stage 2 upper genital tract prolapse indicated for surgery.
* Linked to inflammatory or immune status:

  * With a known hypersensitivity to one of DESIRIAL®'s components (hyaluronic acid, mannitol), to the antiseptic solution, to amide local anesthetics or to one of the components of anesthesia products planned to be used;
  * Presence of clinical signs of inflammation in or close to the area of interest or treatment for these affections;
  * History of or ongoing autoimmune disease.
* Linked to infection:

  * Presence of bacterial, fungal or viral infection in or close to the area of interest or treatment for these affections;
  * With previous history of streptococcal illness (such as recurrent sore throat or acute articular rheumatism);
  * History of Toxic Shock Syndrome.
* Linked to neoplasia:

  * Ongoing or history of cancer in areas close to the injection site (vulvar, vaginal or cervical cancers);
  * Ongoing cancer distant from the injection site. Hormone-dependent breast cancer survivors must be in complete remission after anti-estrogen treatment (tamoxifen, aromatase inhibitor) to be eligible.
* Linked to previous or ongoing treatments:

  * Anti-estrogen treatment (tamoxifen, aromatase inhibitor) for hormone-dependent breast cancer within 1 year prior to inclusion;
  * Treatment with a trophically targeted electromagnetic treatment of the vaginal mucosa (pulsed CO2 laser, LED, radiofrequency, etc.) within 6 months prior to inclusion;
  * Treatment with anticoagulant, antiplatelet agents, NSAIDs or Vitamin C within 1 week prior to inclusion;
  * Local hyaluronic acid-like hydrating treatment within 4 weeks prior to inclusion;
  * Under hormonal treatment: Local vaginal estrogen alone including phytoestrogen, or estrogen-progestogen (rings, creams, ovules, gels) therapy within 1 week prior to inclusion; transdermal estrogen alone or estro-progestogen therapy within 4 weeks prior to inclusion; Tibolone within 4 weeks prior to inclusion; Oral estrogen alone including phytoestrogen, progestogen alone, or estro-progestogen therapy within 8 weeks prior to inclusion; Androgen therapy (including oral or vaginal DHEA) within 8 weeks prior to inclusion; Intrauterine progestogen therapy within 8 weeks prior to inclusion; Progestogen implants or estrogen alone injectable therapy within 3 months prior to inclusion; Estrogen pellet therapy or progestogen injectable therapy within 6 months prior to inclusion;
  * Selective estrogen receptor modulator (SERM) treatment targeted against vaginal dryness (Ospemifene, etc) within 4 weeks prior to inclusion;
  * Antidepressant agents within 4 weeks prior to inclusion;
  * History of vulvovaginal treatment with DESIRIAL® or similar indication implants (resorbable or slowly resorbable) within 1 year prior to inclusion;
  * History of vestibular and/or vaginal treatment with non resorbable implants;
  * Total injection volume of cross-linked hyaluronic acid >19 mL within 1 year prior to inclusion.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
Variation of most bothersome symptom | 12 weeks after Day 0
  Changes in mean Most Bothersome Symptom (MBS) severity score from baseline (Visit 1) to 12 weeks after a single injection of DESIRIAL® in comparison to a placebo (DO group versus PAD group).
  Symptom intensity is assessed using a 4-score scale (from 0 to 3) with minimum score representing a better outcome. Score 0 corresponds to "None", score 1 to "Mild", score 2 to "Moderate" and score 3 to "Severe".

SECONDARY OUTCOMES:
Variation of most bothersome symptom (MBS) | 4 weeks, 12 weeks, 16 weeks, 24 weeks, 36 weeks, 48 weeks and 52 weeks after Day 0
  Changes in mean severity score of MBS after a single injection of DESIRIAL® as detailed:
  * From baseline (V1) to 4 weeks after a single injection of DESIRIAL® in comparison to placebo (DO versus PAD group);
  * From baseline (Visit 1) to 4, 24, 36 and 52 weeks post-injection for patients in DO group;
  * From Visit 3 (12 weeks) to 16, 24, 36 and 48 weeks for patients in PAD group.
  Symptom intensity is assessed using a 4-score scale (from 0 to 3) with minimum score representing a better outcome. Score 0 corresponds to "None", score 1 to "Mild", score 2 to "Moderate" and score 3 to "Severe".
Variation of other moderate to severe symptoms | 4 weeks, 12 weeks, 16 weeks, 24 weeks, 36 weeks, 48 weeks and 52 weeks after Day 0
  Changes in mean severity score of other moderate to severe symptoms after a single injection of DESIRIAL® as detailed:
  * From baseline (Visit 1) to 4 and 12 weeks after a single injection of DESIRIAL® in comparison to placebo (DO versus PAD group);
  * From baseline (Visit 1) to 4, 12, 24, 36 and 52 weeks post-injection for patients in DO group;
  * From Visit 3 (12 weeks) to 16, 24, 36 and 48 weeks for patients in PAD group.
  Symptom intensity is assessed using a 4-score scale (from 0 to 3) with minimum score representing a better outcome. Score 0 corresponds to "None", score 1 to "Mild", score 2 to "Moderate" and score 3 to "Severe".
Percentage of responders | 12 weeks after Day 0
  Percentages of patients with a most bothersome symptom score less than or equal to 1 (mild) at week 12 in comparison to placebo (DO group versus PAD group)
Variation of sexual function | 4 weeks, 12 weeks, 16 weeks, 24 weeks, 36 weeks, 48 weeks and 52 weeks after Day 0
  Changes in Female Sexual Function Index (FSFI) scores after a single DESIRIAL® injection:
  * From baseline (Visit 1) to 4 and 12 weeks after a single injection of DESIRIAL® in comparison to a placebo (DO group versus PAD group);
  * From baseline (Visit 1) to 4, 12, 24, 36 and 52 weeks post-injection for patients in DO group;
  * From Visit 3 at 12 weeks to 16, 24, 36 and 48 weeks for patients in PAD group.
  FSFI consists in 19 questions with multiple-choice responses coded from 0.0 to 5.0. Each score has a specific meaning depending on the question. The scale has six sexual domains. The maximum score for each domain is 6.0, obtained by summing item responses and multiplying by a correction factor. The total composite sexual function score is a sum of domain scores and ranges from 2.0 (not sexually active and no desire) to 36.0.
Variation of vaginal pH | 4 weeks, 12 weeks, 16 weeks, 24 weeks, 36 weeks, 48 weeks and 52 weeks after Day 0
  Changes in pH after a single DESIRIAL® injection:
  * From baseline (Visit 1) to 4 and 12 weeks after a single injection of DESIRIAL® in comparison to a placebo (DO group versus PAD group);
  * From baseline (Visit 1) to 4, 12, 24, 36 and 52 weeks post-injection for patients in DO group;
  * From Visit 3 (12 weeks) to 16, 24, 36 and 48 weeks for patients in PAD group.
Report of adverse events | Through study completion, up to 52 weeks for DO group and up to 48 weeks for PAD group
  Evaluation of product tolerance by collection of adverse events

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (6):
  - Gynecology private office, Antwerp
  - Cabinet Gynécologie Obstétrique, Liège
  - Gynaecologisch Centrum, Mechelen
  - Gynaecologie Dr Deniz Gulcan, Meise
  - Cabinet Dr Ali Bennani, Wavre
  - MIRHA, Zaventem
- France (8):
  - Clinique Georges V, Bordeaux
  - CHRU Jeanne de Flandres, Lille
  - Cabinet de gynécologie, Marseille
  - Cabinet de Gynécologie, Paris
  - Cabinet de gynécologie, Perpignan
  - Polyclinique de l'Atlantique, Saint-Herblain
  - Cabinet de Gynécologie, Tarnos
  - Cabinet de gynécologie, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bensmail H, Marchand Lamiraud F, Martin C, Pelckmans S, Cha'ban F, Siboni Frisch A, Deniz G, Sabban Serfati P, Caubo B, Gurriet B, Petit Breuilh I, Pastijn AI, Berreni N, Cosson M. Hyaluronic acid injection to treat symptoms of vulvovaginal atrophy and improve sexual function in postmenopausal women: A 52-week long-term follow-up. Maturitas. 2025 Oct;201:108687. doi: 10.1016/j.maturitas.2025.108687. Epub 2025 Aug 5. PMID 40773978
- [Derived] Marchand Lamiraud F, Bensmail H, Martin C, Pelckmans S, Cha'ban F, Siboni Frisch A, Deniz G, Sabban Serfati P, Caubo B, Gurriet B, Petit Breuilh I, Pastijn AI, Berreni N, Cosson M. Hyaluronic acid injection to treat symptoms of vulvovaginal atrophy in postmenopausal women: A 12-week randomised, placebo-controlled, multicentric study. Maturitas. 2025 Jun;197:108264. doi: 10.1016/j.maturitas.2025.108264. Epub 2025 Apr 12. PMID 40273666